CLINICAL TRIAL: NCT03877367
Title: Immediate Impact of Extremity Manipulation on an Upper Extremity (UE) Balancing Task
Brief Title: Comparison of Balance Changes After Chiropractic Adjustments in Health Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parker University (Other)
Collaborators: University of Houston (Other); Whittier University (Unknown); University of Miami (Other); Private Practice (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Parker19_03
Record Dates: First submitted 2019-03-13; First posted 2019-03-15 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Postural Balance; Musculoskeletal Manipulation
Keywords: Chiropractic manipulation; Extremity manipulation; Balance task

STUDY DESIGN:
Intervention Model Description: The study will be a patient and outcome assessor blinded, cross-over randomized clinical trial. Participants will randomized into two groups.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Upper Extremity Group, Day 1 (Experimental): Day 1: This group will receive a pre-test, upper extremity intervention, and post-test.
  Day 2: This group will receive a pre-test, lower extremity intervention, and post-test.
  Interventions: Other: Upper extremity manipulation
- Lower Extremity Group, Day 2 (Experimental): Day 1: This group will receive a pre-test, lower extremity intervention, and post-test.
  Day 2: This group will receive a pre-test, upper extremity intervention, and post-test.
  Interventions: Other: Upper extremity manipulation

INTERVENTIONS:
Other: Upper extremity manipulation — An upper extremity (glenohumeral, humeroulnar and radioulnar joints, bilaterally) or a lower extremity (coxofemoral, tibiofemoral, and tibiotalar, bilaterally) manipulation series.
  Other Names: Manipulation

SUMMARY:
This study will examine the effect of upper and lower extremity manipulations on an upper extremity balancing task.

DETAILED DESCRIPTION:
Spinal manipulation has long been thought to have beneficial effects on posture, balance and proprioception; however, only a single study has investigated the effect of chiropractic treatment of the extremities on balance and posture. In a previous study, it was noted that lower extremity manipulation led to more ordered behavior on a dynamic, lower extremity balance task. It was also found that upper extremity manipulation led to less ordered behavior with same lower extremity balance task. Further studies are needed not only to validate this theory, but to further clarify the mechanism regarding specificity of manipulation to task.

ELIGIBILITY:
Inclusion Criteria:

* Between the age 18 years old and 35 years old
* Cleared to be treated in Parker Wellness Clinic

Exclusion Criteria:

* Hx of neurological disorders
* Hx of musculoskeletal disorders/injuries that could impact his/her ability to stand upright
* Currently known to be pregnant
* Compromised vision (beyond the wearing of corrective lenses)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-07-24 (Actual)

PRIMARY OUTCOMES:
Head Sensor to calculate angle of head inclination | 30 seconds
  There will be a sensor placed on each participant's head (in a neoprene headband), as well as on the midpoint of the tube. The head sensor will be used to calculate the angle of head inclination. The sensor on the tube will be used to calculate Sample Entropy as well as general kinematics.

SECONDARY OUTCOMES:
Ground reaction force | less than 1 minute
  Participants will be standing on a force plate that will characterize their ground reaction forces, eyes open without tube (EONT) versus eyes closed without the tube (ECNT).
Center of pressure | less than 1 minute
  Participants will be standing on a force plate that will characterize their center of pressure, EONT versus eye open with the tube horizontally (EOWT).
Velocity to measure sway. | less than 1 minute
  Participants will be standing on a force plate that will characterize their velocity of sway, EOWT versus eye closed with tube held horizontally (ECWT).
Sway: measuring distance | less than 1 minute
  Participants will be standing on a force plate that will characterize their distance of sway, EOWT versus ECWT.
acceleration to measure sway | less than 1 minute
  Participants will be standing on a force plate that will characterize their acceleration of sway, EOWT versus ECWT.

CONTACTS AND LOCATIONS:
Locations (1):
- Parker University, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Malaya CA, Haworth J, Pohlman KA, Smith DL. Immediate impact of extremity manipulation on dual task performance: a randomized, crossover clinical trial. Chiropr Man Therap. 2021 Feb 5;29(1):6. doi: 10.1186/s12998-021-00366-5. PMID 33541378